CLINICAL TRIAL: NCT02016144
Title: Optimal Length of the Pre-inserted Endotracheal Tube for Obtaining Good View of Laryngeal Opening for Nasal Fibreoptic Intubation
Brief Title: Optimal Length of Pre-inserted ETT for Nasal Fiber Optic Intubation
Status: Completed | Type: Observational
Sponsor: Seoul National University Dental Hospital (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Assistant professor, Seoul National University Dental Hospital
Other Study IDs: JLee_optimal_length
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Nasal Fiberoptic Intubation
Keywords: Airway management; Fiber optic technology; Intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is intended to find the optimal length of pre-inserted ETT for nasal fiberoptic intubation and the equation to predict it.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* aged 20-65 yr (adults)

Exclusion Criteria:

* rhinitis
* bleeding diatheses
* requirement of awake intubation
* a previous major oral and maxillofacial surgery history
* anatomical deformity of the face, neck and upper airway

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo an elective oral and maxillofacial surgery requiring a nasal intubation of ETT for general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
optimal length of pre-inserted ETT for nasal fiberoptic intubation | during endotracheal intubation for general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D, Principal Investigator — Seoul National University Dental Hospital
Locations (1):
- Seoul National University Dental Hospital, Seoul, South Korea